CLINICAL TRIAL: NCT01291251
Title: Compliance With Antibiotic Treatment in General Practice
Status: Completed | Type: Observational
Sponsor: Norwegian Medical Association (Other)
Responsible Party: Principal Investigator, Torunn Bjerve Eide, MD, Norwegian Medical Association
Other Study IDs: VH-TBE-1
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The guidelines of The Norwegian authorities concerning the use of antibiotics in general practice state that for several common diseases such as pneumonia and tonsillitis, antibiotics should be given four times daily instead of three times daily. The study´s aim is to see whether the patient compliance is significantly reduced in antibiotic regimes of 3 or 4 daily doses as compared to 1 or 2 daily doses.

DETAILED DESCRIPTION:
All patients given antibiotic tablets, independent of diagnosis and medicament, are included. All patients give a written consent. Within a week after the end of the treatment all patients are contacted by one of the authors and asked a few standardized questions concerning their compliance with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any patient given antibiotics for any cause

Exclusion Criteria:

* Use of mixture instead of tablets
* Tablets administrated by public health care services

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in two different primary care clinics.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mette Brekke, Ph D, Study Director — University of Oslo
Locations (2):
- Norway (2):
  - Hisøy legekontor, Arendal, Aust-Agder
  - Froland legekontor, Frøland, Aust-Agder